CLINICAL TRIAL: NCT05368103
Title: A Phase 2A, Open Label, Proof of Concept Trial of Daxdilimab for the Treatment of Moderate To Severe Alopecia Areata
Brief Title: Study of DAXDILIMAB for the Treatment of Moderate-to-Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-DAX-201
Record Dates: First submitted 2022-04-11; First posted 2022-05-10 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daxdilimab (Experimental): Nine sets of Daxdilimab injections over a total of 32 weeks.
  Interventions: Biological: Daxdilimab

INTERVENTIONS:
Biological: Daxdilimab — Daxdilimab will be administered subcutaneously as two injections for each dose.
  Other Names: HZN-7734

SUMMARY:
The purpose of this study is to assess the preliminary efficacy, safety, tolerability, PK, and PD of Daxdilimab in participants with moderate to severe AA, with ≥50% and ≤95% total scalp hair loss as defined by the SALT score at Screening and Day 1.

DETAILED DESCRIPTION:
Approximately 30 participants will be enrolled to receive daxdilimab administered subcutaneously over 32 weeks. The maximum trial duration per participant is approximately 52 weeks, including up to 30 days for the screening period, 32 weeks for the open-label treatment period where participants will receive daxdilimab and approximately 16 weeks for the follow-up period. Safety evaluations will be performed regularly throughout the course of the study.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.
3. Adult men or women 18 to 65 years of age.
4. Willing to keep the same hair style and color (eg, hair products, process, and timing for hair appointments) for the duration of the trial.
5. Clinical diagnosis of moderate-to-severe AA - defined as meeting the following criteria:

   * Presence of ≥ 50% and ≤ 95% total scalp hair loss at screening and baseline (Day 1) defined by the SALT score.
   * Duration of current episode of hair loss >3 months but <7 years at screening and Day 1, along with investigators' assessment that hair regrowth is possible.
   * No evidence of active regrowth present at baseline and no known history of significant regrowth, as per investigator's judgement, over the last 6 months.

Exclusion Criteria:

1. Individuals involved in the conduct of the trial, their employees, or immediate family members of such individuals.
2. Any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with the evaluation of the IP or interpretation of trial results.
3. History of allergy, hypersensitivity reaction, or anaphylaxis to any component of the IP or to a previous monoclonal antibody (mAb) or human immunoglobulin (Ig) therapy.
4. Participant has had excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths within 4 weeks prior to Day 1 or is not willing to minimize natural and artificial sunlight exposure during the trial. Use of sunscreen products and protective apparel are recommended when sun exposure cannot be avoided.
5. Known history of a primary immunodeficiency or an underlying condition such as known human immunodeficiency virus (HIV) infection, a positive result for HIV infection, splenectomy, or any underlying condition that in the opinion of the investigator significantly predisposes the participant to infection.
6. Confirmed positive test for hepatitis B serology defined as:

   * Hepatitis B surface antigen (HBsAg), or
   * Hepatitis B core antibody (HBcAb or anti-HBc)
7. Positive test for hepatitis C virus antibody.
8. Active tuberculosis (TB), or a positive TB test at Screening. Participant will be evaluated for latent TB infection with a purified protein derivative (PPD) test or a QuantiFERON-TB Gold test. Participants who demonstrate evidence of latent TB infection (either PPD ≥5 mm of induration or positive QuantiFERON-TB Gold test, irrespective of bacille Calmette-Guérin vaccination status will not be allowed to participate in the trial, unless documented history of appropriate treatment for active or latent TB. Participants with an indeterminate test result can repeat the test, but if the repeat test is also indeterminate, they are excluded.
9. Any severe herpes virus family infection (including Epstein-Barr virus, cytomegalovirus [CMV]) at any time prior to Day 1, including, but not limited to, disseminated herpes, herpes encephalitis, recent recurrent herpes zoster (defined as 2 episodes within the last 2 years), or ophthalmic herpes.
10. Any herpes zoster, CMV, or Epstein-Barr virus infection that was not completely resolved 12 weeks prior to Day 1.
11. Any of the following within 30 days prior to signing the ICF and though Day 1:

    * Clinically significant active infection in the opinion of the investigator, including ongoing, and chronic infection requiring antibiotics or antiviral medication (chronic nail infections are allowed). Note: Participant with a limited recurrence of a cold sore or herpes genitalis between ICF signature and Day 1 could be eligible based on the investigator's judgement.
    * Any infection requiring hospitalization or treatment with intravenous (IV) anti-infectives.
    * A participant with a documented positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test may be rescreened at least 2 weeks after a positive test if the participant is asymptomatic and at least 3 weeks after resolution of symptomatic Coronavirus Disease 2019 (COVID-19) illness.
12. Opportunistic infection requiring hospitalization or parenteral antimicrobial treatment within 2 years prior to Day 1.
13. Any acute illness or evidence of clinically significant active infection, such as fever ≥ 38.0°C (≥ 100.5°F) on Day 1.
14. History of clinically significant cardiac disease including unstable angina; myocardial infarction within 6 months prior to Day 1; congestive heart failure; arrhythmia requiring active therapy, except for clinically insignificant extra systoles, or minor conduction abnormalities; or presence of clinically significant abnormality on ECG if, in the opinion of the investigator, it would increase the risk of trial participation.
15. History of cancer or lymphoproliferative disease within 5 years prior to Day 1, except as follows:

    * In situ carcinoma of the cervix treated with apparent success with curative therapy > 12 months prior to Screening, or
    * Nonmetastatic cutaneous basal cell or squamous cell carcinoma of the skin treated with apparent success with curative therapy.
16. Active forms of other inflammatory skin disease(s) or evidence of other skin conditions (eg, psoriasis, seborrheic dermatitis, lupus) at the time of the Screening and through Day 1, that in the opinion of the investigator might interfere with evaluation of AA and the assessment of the activity measures.
17. Presence of another form of alopecia (except for androgenic alopecia).
18. History of male or female pattern hair loss > Hamilton stage III or > Ludwig stage II.
19. History or presence of hair transplants.
20. History or presence of micropigmentation of the scalp (Note: microblading of the eyebrows is permitted).
21. Use of steroids (systemic and intralesional), anthralin, squaric acid, diphenylcycloprophenone (DPCP), dinitrochlorobenzene (DCNB), protopic, minoxidil, or any other medication which in the opinion of the investigator may affect hair regrowth within 4 weeks of Day 1 visit. Note: Intranasal and inhaled corticosteroids are allowed, eye and ear drops containing corticosteroids are also allowed.
22. Use of platelet-rich plasma injections in the last 12 weeks prior to Day 1.
23. Topical medicated treatment that could affect AA including, but not limited to, topical corticosteroids, calcineurin inhibitors, antimicrobials, medical devices within 2 weeks of Day 1 visit. Note: Topical corticosteroids are permitted outside of the scalp, eyebrows, and eyelids.
24. Participants who have had previous treatment with any biologic B-cell-depleting therapy (eg, rituximab, ocrelizumab, or ofatumumab) or other B-cell targeting therapy (eg, belimumab) within 12 months before Day 1.
25. Participants who have received previous treatment with pDC inhibiting therapies (eg, anti-ILT7, anti-blood dendritic cell antigen 2 [BDCA2]).
26. Inadequate response to adequate trial of oral Janus Kinase (JAK) inhibitors. Previous exposure to topical JAK inhibitors is acceptable, regardless of response.
27. Any biologic or conventional disease-modifying antirheumatic drugs (DMARD), immunosuppressant (eg, cyclosporine, methotrexate, or azathioprine), JAK-inhibitors, interferon (IFN) blocking therapies, or antiproliferative agents, if last dose was taken: a. within 8 weeks prior to Day 1 or b. drug-specific 5 half-lives elimination period (if longer than 8 weeks).
28. Participant has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
29. Currently receiving a nonbiological IP or device or has received one within 4 weeks prior to Day 1 or within 5 published half-lives, whichever is longer.
30. Participant has received any ultraviolet (UV)-B phototherapy (including tanning beds), has had psoralen-UV-A (PUVA) treatment, or excimer laser within 4 weeks prior to Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (6):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - First OC Dermatology Research, Inc., Fountain Valley, California
  - ForCare Clinical Research, Tampa, Florida
  - DS Research, Louisville, Kentucky
  - Progressive Clinical Research, P.A., San Antonio, Texas
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (7):
  - Enverus Medical Research, Surrey, British Columbia
  - Dr Dusan Sajic Medicine Professional Corporation, Guelph, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Innovaderm Research, Montreal, Quebec
  - Centre de Recherche Saint-Louis (Quebec), Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 participants were enrolled at 5 trial centers located in the United States and 7 trial centers in Canada between 27 April 2022 and 26 January 2024.
Pre-assignment Details: Of the 55 participants who were screened for enrolment in the trial, 25 were screen failures. A total of 30 participants were enrolled and received daxdilimab.
Groups:
- Daxdilimab 300 mg: Participants received 300 mg daxdilimab as two subcutaneous (SC) injections every 4 weeks (Q4W) for 32 weeks. Participants were followed-up until Week 48.
Period: Overall Study
Arm/Group | Daxdilimab 300 mg
Started | 30
Received Daxdilimab | 30
Completed | 22
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6
  Black or African American | 2
  White | 20
  Other | 2
Severity of Alopecia Tool (SALT) Score [Mean (Standard Deviation); unit: score on a scale] — The SALT score determined the degree of hair loss based on the percentage of scalp surface area involved on the top, back, and each side of the scalp for alopecia areata (AA). The Investigator determined the percent scalp hair loss in a given quadrant, multiplied this by the total scalp area delineated by that quadrant, and summed the resultant numbers for each quadrant to give the total percent scalp hair loss with a range of 0-100.
  score on a scale | 74.4 (15.72)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in SALT Score at Week 24
Description: The SALT score determined the degree of hair loss based on the percentage of scalp surface area involved on the top, back, and each side of the scalp for AA. The Investigator determined the percent scalp hair loss in a given quadrant, multiplied this by the total scalp area delineated by that quadrant, and summed the resultant numbers for each quadrant to give the total percent scalp hair loss with a range of 0-100. Higher scores indicated more severe AA symptoms. A decrease in SALT score from baseline indicated a reduction in AA symptoms.
  Baseline indicates last non-missing valid observation prior to the first dose of daxdilimab.
Time Frame: Baseline to Week 24
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Mean (Standard Deviation); unit: percent change in score on a scale
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent change in score on a scale | -12.6 (35.15)

2. Secondary Outcome: Percent Change From Baseline in SALT Score at Weeks 12, 16, 20, 28, 32, and 36
Description: as for outcome 1
Time Frame: Baseline to Weeks 12, 16, 20, 28, 32, and 36
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Mean (Standard Deviation); unit: percent change in score on a scale
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent change in score on a scale
  Week 12 | -5.4 (21.57)
  Week 16 | -8.1 (26.58)
  Week 20 | -10.0 (30.10)
  Week 28 | -16.2 (34.35)
  Week 32 | -17.2 (37.16)
  Week 36 | -18.2 (37.22)

3. Secondary Outcome: Percentage of Participants Who Achieved a ≥ 50% Reduction in SALT Score From Baseline at Weeks 12, 16, 20, 24, 28, 32, and 36
Description: as for outcome 1
Time Frame: Baseline to Weeks 12, 16, 20, 24, 28, 32, and 36
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 12 | 3.3 [0.1 to 17.2]
  Week 16 | 10.0 [2.1 to 26.5]
  Week 20 | 13.3 [3.8 to 30.7]
  Week 24 | 20.0 [7.7 to 38.6]
  Week 28 | 20.0 [7.7 to 38.6]
  Week 32 | 20.0 [7.7 to 38.6]
  Week 36 | 20.0 [7.7 to 38.6]

4. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 10 at Weeks 12, 16, 20, 24, 28, 32, and 36
Description: The SALT score determined the degree of hair loss based on the percentage of scalp surface area involved on the top, back, and each side of the scalp for AA. The Investigator determined the percent scalp hair loss in a given quadrant, multiplied this by the total scalp area delineated by that quadrant, and summed the resultant numbers for each quadrant to give the total percent scalp hair loss with a range of 0-100. Higher scores indicated more severe AA symptoms.
  Baseline indicates last non-missing valid observation prior to the first dose of daxdilimab.
Time Frame: Weeks 12, 16, 20, 24, 28, 32, and 36
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 12 | 0.0 [0.0 to 11.6]
  Week 16 | 0.0 [0.0 to 11.6]
  Week 20 | 0.0 [0.0 to 11.6]
  Week 24 | 3.3 [0.1 to 17.2]
  Week 28 | 6.7 [0.8 to 22.1]
  Week 32 | 10.0 [2.1 to 26.5]
  Week 36 | 13.3 [3.8 to 30.7]

5. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 20 at Weeks 12, 16, 20, 24, 28, 32, and 36
Description: as for outcome 4
Time Frame: Weeks 12, 16, 20, 24, 28, 32, and 36
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 12 | 0.0 [0.0 to 11.6]
  Week 16 | 0.0 [0.0 to 11.6]
  Week 20 | 6.7 [0.8 to 22.1]
  Week 24 | 13.3 [3.8 to 30.7]
  Week 28 | 16.7 [5.6 to 34.7]
  Week 32 | 16.7 [5.6 to 34.7]
  Week 36 | 16.7 [5.6 to 34.7]

6. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 30 at Weeks 12, 16, 20, 24, 28, 32, and 36
Description: as for outcome 4
Time Frame: Weeks 12, 16, 20, 24, 28, 32, and 36
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 12 | 6.7 [0.8 to 22.1]
  Week 16 | 10.0 [2.1 to 26.5]
  Week 20 | 10.0 [2.1 to 26.5]
  Week 24 | 16.7 [5.6 to 34.7]
  Week 28 | 16.7 [5.6 to 34.7]
  Week 32 | 16.7 [5.6 to 34.7]
  Week 36 | 20.0 [7.7 to 38.6]

7. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 50 at Weeks 12, 16, 20, 24, 28, 32, and 36
Description: as for outcome 4
Time Frame: Weeks 12, 16, 20, 24, 28, 32, and 36
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 12 | 16.7 [5.6 to 34.7]
  Week 16 | 23.3 [9.9 to 42.3]
  Week 20 | 26.7 [12.3 to 45.9]
  Week 24 | 26.7 [12.3 to 45.9]
  Week 28 | 30.0 [14.7 to 49.4]
  Week 32 | 30.0 [14.7 to 49.4]
  Week 36 | 30.0 [14.7 to 49.4]

8. Secondary Outcome: Percent Change From Baseline in SALT Score at Weeks 40, 44, and 48
Description: as for outcome 1
Time Frame: Baseline to Weeks 40, 44, and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Mean (Standard Deviation); unit: percent change in score on a scale
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent change in score on a scale
  Week 40 | -19.4 (37.72)
  Week 44 | -20.6 (40.67)
  Week 48 | -22.1 (41.43)

9. Secondary Outcome: Percentage of Participants Who Achieved a ≥ 50% Reduction in SALT Score From Baseline at Weeks 40, 44, and 48
Description: as for outcome 1
Time Frame: Baseline to Weeks 40, 44, and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 40 | 20.0 [7.7 to 38.6]
  Week 44 | 26.7 [12.3 to 45.9]
  Week 48 | 23.3 [9.9 to 42.3]

10. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 10 at Weeks 40, 44 and 48
Description: as for outcome 4
Time Frame: Weeks 40, 44 and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 40 | 10.0 [2.1 to 26.5]
  Week 44 | 10.0 [2.1 to 26.5]
  Week 48 | 13.3 [3.8 to 30.7]

11. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 20 at Weeks 40, 44 and 48
Description: as for outcome 4
Time Frame: Weeks 40, 44 and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 40 | 16.7 [5.6 to 34.7]
  Week 44 | 16.7 [5.6 to 34.7]
  Week 48 | 16.7 [5.6 to 34.7]

12. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 30 at Weeks 40, 44 and 48
Description: as for outcome 4
Time Frame: Weeks 40, 44 and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 40 | 20.0 [7.7 to 38.6]
  Week 44 | 20.0 [7.7 to 38.6]
  Week 48 | 16.7 [5.6 to 34.7]

13. Secondary Outcome: Percentage of Participants Who Had an Absolute SALT Score ≤ 50 at Weeks 40, 44 and 48
Description: as for outcome 4
Time Frame: Weeks 40, 44 and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent of participants
  Week 40 | 26.7 [12.3 to 45.9]
  Week 44 | 30.0 [14.7 to 49.4]
  Week 48 | 23.3 [9.9 to 42.3]

14. Secondary Outcome: Serum Concentration of Daxdilimab
Description: Blood samples were collected at the visits and time points specified.
  All post-baseline concentrations below the limit of quantification (BLQ) were imputed as half of the lower limit of quantification value.
Time Frame: Baseline: 2 hours post-dose; Weeks 4-32: Pre-dose; Weeks 36-48: Any time during the visit.
Population: Pharmacokinetic (PK) Analysis Set: Included all participants who received any dose of daxdilimab and had at least one measurable PK concentration post-dose. Only participants with evaluable data at each timepoint were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
ng/mL
  Baseline | 0.640 (1.354)
  Week 4 | 6.698 (3.514)
  Week 8 | 8.823 (4.439)
  Week 12: number analyzed (Participants) | 28
  Week 12 | 9.978 (5.569)
  Week 16: number analyzed (Participants) | 27
  Week 16 | 9.582 (5.410)
  Week 20: number analyzed (Participants) | 27
  Week 20 | 9.473 (5.616)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 10.322 (6.154)
  Week 28: number analyzed (Participants) | 24
  Week 28 | 10.595 (6.663)
  Week 32: number analyzed (Participants) | 25
  Week 32 | 10.638 (6.549)
  Week 36: number analyzed (Participants) | 25
  Week 36 | 10.480 (6.074)
  Week 40: number analyzed (Participants) | 25
  Week 40 | 3.543 (2.878)
  Week 44: number analyzed (Participants) | 22
  Week 44 | 1.309 (1.218)
  Week 48: number analyzed (Participants) | 22
  Week 48 | 0.430 (0.465)

15. Secondary Outcome: Percent Change From Baseline in Plasmacytoid Dendritic Cell (pDC) Levels
Description: Blood samples were collected at the visits and timepoints specified and analyzed using flow cytometry.
Time Frame: Baseline to Weeks 4, 12, 24, 32, 36 and 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab. Only participants with evaluable data at each time point were included.
Measure: Median (Full Range); unit: percent change in pDC levels
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
percent change in pDC levels
  Week 4: number analyzed (Participants) | 23
  Week 4 | -88.89 [-100 to -16.7]
  Week 12: number analyzed (Participants) | 21
  Week 12 | -87.50 [-100 to 33.3]
  Week 24: number analyzed (Participants) | 18
  Week 24 | -85.71 [-100 to -50]
  Week 32: number analyzed (Participants) | 18
  Week 32 | -85.71 [-100 to 33.3]
  Week 36: number analyzed (Participants) | 18
  Week 36 | -82.86 [-96.6 to 66.7]
  Week 48 | -40.00 [-90.5 to 200]

16. Secondary Outcome: Number of Participants Who Experienced an Anti-drug Antibody (ADA) Response
Description: The number of participants who experienced an ADA response was defined as participants with ADA positive post-baseline only or boosted their preexisting ADA during the study.
Time Frame: Baseline and Weeks 4, 8, 12, 24, and 36: Pre-dose
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
Participants | 1

17. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was any untoward medical occurrence in a participant that was not present prior to treatment but appeared following treatment, was present at treatment initiation but worsened during treatment, or was present at the treatment initiation but resolved and then reappeared while the participant was on treatment and did not necessarily have a causal relationship with the treatment.
  A serious TEAE was defined as any medical occurrence that had any of the following consequences:
  * Resulted in death.
  * Was life-threatening.
  * Required in-patient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent or significant disability/incapacity.
  * Was a congenital anomaly/birth defect.
Time Frame: Day 1 to Week 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
Participants
  TEAEs | 23
  Serious TEAEs | 0

18. Secondary Outcome: Number of Participants Who Experienced an Adverse Event of Special Interest (AESI)
Description: An AESI was defined as a serious or non-serious adverse event of scientific and medical interest specific to understanding the treatment and may have required close monitoring and collection of additional information by the investigator.
  The following were defined as AESIs:
  * Hypersensitivity reaction, including anaphylaxis.
  * Severe viral infection/reactivation.
  * Opportunistic infection.
  * Malignancy (except non-melanoma skin cancer).
Time Frame: Day 1 to Week 48
Population: Safety Analysis Set: Included all participants who received any dose of daxdilimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Daxdilimab 300 mg
Number analyzed (Participants) | 30
Participants | 2

ADVERSE EVENTS:
Time Frame: Day 1 to Week 48
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of daxdilimab.
Arm/Group | Daxdilimab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 17/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daxdilimab 300 mg (N=30)
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Injection site reaction (General disorders) | 6
Seasonal allergy (Immune system disorders) | 2
COVID-19 (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT05368103/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT05368103/SAP_001.pdf